CLINICAL TRIAL: NCT05306197
Title: Improving Performance of Combat Soldiers by Utilizing Attentional Training Based on Eye Tracking - Improvement of Combat Performance
Brief Title: Improving Performance of Combat Soldiers by Utilizing Attentional Training Based on Eye Tracking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to deteriorating operative and security conditions in the country, we were unable to continue meeting with the troops for data collection.
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TAU-GCFTperformance
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Military Combat Performance
Keywords: Attention Bias Modification; Randomized Control Trial; Eye-tracking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gaze-Contingent Feedback Training (toward threat) (Experimental): In the task, 30 different matrices, each consisting of 16 faces, will be presented. Each matrix includes 8 angry faces and 8 neutral, 8 women and 8 men, and the locations are counterbalanced between matrices. The participants are asked to view the matrices in any way they choose, and the eye-tracking camera records their viewing location relative to the stimuli presented on the screen. At the beginning of each training session, the soldier will choose to which music he would like to listen during the 12-minute session from a diverse list of music. After calibrating the eye-tracker, the participant will be instructed to view matrices of faces as he chooses, as described above in the assessment task. The music chosen by the participant will play only when he is looking at threatening faces and it will stop when he looks at neutral faces. Thus, a change in viewing patterns is expected by implementing operant conditioning principles.
  Interventions: Behavioral: Gaze-Contingent Feedback Training
- Active Comparator: RT-Based Attention Bias Modification (toward threat) (Active Comparator): A dot-probe task of 160 trials. Trials begins with a fixation cross (+), on which the participant is asked to focus (500ms). Then two face stimuli (one angry one neutral) are presented above and below the fixation cross (500ms). After the stimuli disappear, a target probe (right- or left-pointing arrowhead) appears in place of one of the face stimuli. The participant is asked to indicate which target probe was presented using a predetermined key. The target probe will remain on the screen until response, after which a new trial will begin.
  Participants are instructed to identify the probe type as quickly and accurately as possible.
  In the training task, all of the target probes will appear in the threat location (angry face). Thus, over multiple trials, learning is expected to occurs such that the threatening face predicts the location of the target probe, thereby achieving the desired change in attention pattern.
  Interventions: Behavioral: Attention Bias Modification
- Non-Contingent Feedback Training (Placebo Comparator): This condition is also based on the eye-tracking task (see Experimental Arm) with a fundamental change - The music chosen by the soldier will play continuously without any reinforcement for looking at threat or neutral faces.
  Interventions: Behavioral: Non-Contingent Feedback Training

INTERVENTIONS:
Behavioral: Gaze-Contingent Feedback Training — Feedback according to participants' viewing patterns, in order to modify their attention toward threat stimuli.
  Arms: Gaze-Contingent Feedback Training (toward threat)
Behavioral: Attention Bias Modification — Attention training via repeated trials of a dot-probe task intended to direct attention toward threat stimuli using threat and neutral face stimuli.
  Arms: Active Comparator: RT-Based Attention Bias Modification (toward threat)
Behavioral: Non-Contingent Feedback Training — Participants listen to a musical track they chose with no operant conditioning.
  Arms: Non-Contingent Feedback Training

SUMMARY:
Military service in combat units entails exposure to traumatic events that require mental adjustment. To develop and efficiently apply attentional interventions aimed at enhancing soldiers' combat performance, it is essential to extensively investigate the efficiency of these training programs, which has yet to been done. The prupose of the current study is to examine the efficiency of the new attention eye-tracking based training, in comparison to RT-based training and to a control group, in improving performance of combat soldiers. In addition, the influence of the attention training on aspects of psychological resilience will also be examined in questionnaires.

DETAILED DESCRIPTION:
Following the explanation to participants regarding the study process, those who give written consent to participate will be randomly placed into one of three groups: GCFT (N=60), ABMT (N=60), and a neutral control group - task based on eye-tracking (N=60). The study will include 2 measurement points during the military service: before the attention training and after the attention training. In each measurement point, the soldiers will complete computerized tasks to measure threat attention, questionnaires, and performance data from shooting ranges and combat fitness.

ELIGIBILITY:
Inclusion Criteria:

* Each soldier from the cohort that will give his written consent will be able to participate in the study.

Exclusion Criteria:

* Hebrew proficiency is insufficient to complete the study questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Change in Combat Performance | Approximately 3 months after baseline
  Composite scores for Static marksmanship, simulator shooting performance (Bagira), running test grades, and obstacle course grades will be gathered from soldiers' commanders before and after intervention sessions to test for change.

SECONDARY OUTCOMES:
Post-Combat Trauma | Change from baseline Post-Combat PTSD Symptoms at approximately 3 months
  Score on on self-report questionnaire Posttraumatic stress disorder checklist for DSM-5 (PCL-5). The total score, ranging from 0 to 80, reflects PTSD symptom severity, with higher scores representing greater severity.
Post-Combat General Anxiety | Change from baseline Post-Combat General Anxiety Symptoms at approximately 3 months
  Score on self-report questionnaire Generalized Anxiety Disorder questionnaire (GAD-7). The total score, ranging from 0 to 21, reflects GAD symptom severity, with higher scores representing greater severity.
Post-Combat Depression | Change from baseline Post-Combat Depression Symptoms at approximately 3 months
  Score on self-report Patient Health Questionnaire 9 (PHQ-9). The total score, ranging from 0-27, reflects severity of depressive symptoms, with higher scores representing greater severity.

OTHER OUTCOMES:
Post-Training RT-based Attention Bias toward threat | Change from baseline Attention Bias within 3 months of baseline measurement
  Change in Attention Bias will be assessed with a response-time based dot-probe task.
Post-Training Subjective Attention Bias toward threat | Change from baseline Attention Bias within 3 months of baseline measurement
  Change in Subjective Attention Bias will be assessed with a self-reported attention bias using the Attention Bias Questionnaire (ABQ). The total score, ranging from 0 to 36, represents threat-related attention bias, with higher scores representing greater bias toward threat.
Post-Training Eye-tracking Attention Bias toward threat | Change from baseline Attention Bias within 3 months of baseline measurement
  Change in Attention Bias will also be assessed with an eye-tracking task.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wald I, Fruchter E, Ginat K, Stolin E, Dagan D, Bliese PD, Quartana PJ, Sipos ML, Pine DS, Bar-Haim Y. Selective prevention of combat-related post-traumatic stress disorder using attention bias modification training: a randomized controlled trial. Psychol Med. 2016 Sep;46(12):2627-36. doi: 10.1017/S0033291716000945. Epub 2016 Jul 5. PMID 27377418